CLINICAL TRIAL: NCT05028985
Title: A Cohort Study of Early Chronic Obstructive Pulmonary Disease for China Pulmonary Health Study Stage II
Brief Title: Early COPD for China Pulmonary Health Study Stage II
Acronym: EC-CPHS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Capital Medical University (Other); Peking University Third Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Chen Wang, Study Chair, China-Japan Friendship Hospital
Other Study IDs: 82090011
Record Dates: First submitted 2021-06-03; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lung tissues, serum, bronchoalveolar lavage fluid, bronchial epithelial cells, sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early COPD patients: younger than 50 years with 10 or more pack-years smoking history and any of these abnormalities: 1) early airflow limitation (post-bronchodilator forced expiratory volume in the first second(FEV1)/forced vital capacity(FVC) < lower limit of normal), 2) compatible CT abnormalities, 3) rapid decline in FEV1 (≥60 ml/yr).
- Healthy people: healthy without any disabling, physical, neurological, or mental disease and were excluded living in a nursing home.

SUMMARY:
Discovery of the pathogenesis and targets in the progression of early chronic obstructive pulmonary disease

DETAILED DESCRIPTION:
This project is aimed to investigate and explore the heterogeneity during the progression of Chronic Obstructive Pulmonary Disease (COPD) in the early stage, utilizing the large-scale population cohort databases (including "China Pulmonary Health study", "The Cohort Study for Chronic Obstructive Pulmonary Disease in China" and "Acute Exacerbation of COPD Patient Registry in China" ), biological sample libraries(including blood, sputum, expiratory air, bronchoalveolar lavage fluid(BALF), and lung tissue from COPD patients with different stages and phenotypes), and multi-omics sequencing (including scRNA-seq, metabolomics, proteomics, and metagenome). We propose to establish a new standard for COPD stages and subtypes. By analyzing and mining the multi-omics data, it is expected to illustrate the association between clinical phenotype and molecular, cellular and tissue heterogeneities, thus reveal biomarkers related to the progression, clinical phenotypes, and prognosis of early-stage COPD disease.In addition, we will construct different types and stages of COPD animal models for further mechanism studies, such as the different pathogenic factors, innate and adaptive immunity, and the airway microbial ecosystem, so that we can discovered more potential therapeutic target for early-stage COPD. This project can bring a new insight and scientific evidence for COPD treatment.

ELIGIBILITY:
Inclusion Criteria:

* younger than 50 years
* smoking more than 10 pack-years
* early airflow limitation(post-bronchodilator FEV1/FVC< lower limit of normal)

Exclusion Criteria:

* cancer
* other respiratory diseases
* mental illness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: early COPD patients and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
FEV1 annual decline in clinical practice | 2021.1-2024.12
  FEV1 measured by portable spirometry can reflect the progression of early COPD.

SECONDARY OUTCOMES:
dyspnea symptoms | 2021.1-2024.12
  Severity of dyspnea is positively correlated with COPD severity.
frequency of COPD acute exacerbation | 2021.1-2024.12
  The frequency of COPD acute exacerbation refers to the number of acute exacerbations per year.
chest imaging changes | 2021.1-2024.12
  Emphysema and obstruction in small airway will be evaluated by chest computed tomography(CT).
systemic complications | 2021.1-2024.12
  Whether there are systemic complications is related to the prognosis of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wang, Study Chair — Institue of Basic Medical Sciences Chinese Academy of Medical Sciences; Ting Yang, Principal Investigator — China-Japan Friendship Hospital; Jing Wang, Principal Investigator — Institue of Basic Medical Sciences Chinese Academy of Medical Sciences; Huahao Shen, Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine; Wei Wang, Principal Investigator — Capital Medical University; Yahong Chen, Principal Investigator — Peking University Third Hospital; Weining Xiong, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (6):
- China (6):
  - Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Capital Medical University, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Institue of Basic Medical Sciences Chinese Academy of Medical Sciences, Beijing
  - Peking University Third Hospital, Beijing
  - Shanghai Ninth People's Hospital, Shanghai JiaoTong university school of medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No